CLINICAL TRIAL: NCT02494999
Title: A Randomized, Double-blind, Parallel-Controlled Phase III Clinical Trial of a 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants
Brief Title: A Phase III Clinical Trial of a 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JSVCT022
Record Dates: First submitted 2015-07-06; First posted 2015-07-13 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Pneumonia
Keywords: pneumococcal conjugate vaccine; immunogenicity; safety
MeSH Terms: conditions — Pneumonia | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 13-valent pneumococcal conjugate vaccine (Experimental): Single 0.5 ml dose will be given via intramuscular injection in Month 0,2,4 and 10
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine
- Prevnar 13 (Active Comparator): Single 0.5 ml dose will be given via intramuscular injection in Month 0,2,4 and 10
  Interventions: Biological: Prevnar 13

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — 0.5ml vaccine produced by Beijing Minhai Biotechnology Co., Ltd.,three doses with 2 month interval, a booster dose 10 months after the first dose
  Arms: 13-valent pneumococcal conjugate vaccine
Biological: Prevnar 13 — 0.5ml vaccine produced by Wyeth,three doses with 2 month interval, a booster dose 10 months after the first dose
  Arms: Prevnar 13

SUMMARY:
In order to evaluate immunogenicity and safety of a 13-valent pneumococcal conjugate vaccine produced by Beijing Minhai Biotechnology Co., Ltd., a randomized, double-blind, parallel-controlled phase III clinical trial is planned to conduct in healthy infants aged 2 months in China.

DETAILED DESCRIPTION:
There will be two arms. 1200 healthy infants aged 2 months will be randomly assigned (1:1) to receive an experimental vaccine or a comparator vaccine in Month 0,2 and 4 (primary vaccination). All of them will receive a fourth dose as booster vaccination in Month 10.

ELIGIBILITY:
Inclusion Criteria:

* Aged 42-77 days old on the day of inclusion
* Subjects' legal guardians are able to understand and sign the informed consent
* Subjects' legal guardians can and will comply with the requirements of the protocol
* Subjects with temperature <=37.0°C on axillary setting

Exclusion Criteria for First Vaccination:

* Preterm infants or low birth weight infants
* Any administration history of pneumococcal polysaccharide vaccine or pneumococcal conjugate vaccine
* A medical history of culture-confirmed invasive disease caused by Streptococcus pneumonia
* Subject who has allergic history or serious adverse reaction history after vaccination such as allergies, hives, difficulty in breathing, angioedema or abdominal pain
* Subject with congenital malformation, developmental disorder, genetic defects or severe malnutrition
* Subject with epilepsy, a history of seizures or convulsions, or a family history of mental illness
* Known or suspected immune deficiency or immune suppression
* Diagnosed coagulation abnormalities (such as clotting factor deficiency, coagulation disorders, platelet disorder) or significant bruising or blood clotting disorder
* Had immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (not including allergic rhinitis corticosteroid spray treatment, acute uncomplicated dermatitis surfaces corticosteroid therapy) in the past 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of any attenuated live vaccine in last 14 days
* Any prior administration of subunit or inactivated vaccines in last 7 days
* Any acute infection or serious infection needing systemic antibiotics or antiviral treatment in last 7 days
* Any fever with temperature >=38.0°C on axillary setting in last 3 days
* Any other factors judged by investigator, that may interfere subject's compliance with the protocol

Exclusion Criteria for Second/Third and Booster Vaccination:

If one of the following (1) to (3) adverse events (AE) occurs, further vaccination is prohibited, but other study steps can be continued according to the judgment of the investigators; If one of the following (4) to (5) adverse events occurs, the investigator shall determine whether to continue the following vaccination. In the event of one of the following adverse events (6) to (7), vaccination may be postponed within the time window specified in the protocol.

* （1）The subjects have suffered from severe adverse events caused by the previous vaccination.
* （2）The subjects suffered from severe allergic reactions or hypersensitivity after the previous vaccination.
* （3）Known or suspected autoimmune diseases or immunodeficiency diseases，including HIV infection.
* （4）The occurrence of acute or emerging chronic diseases at the time of vaccination.
* （5）Other reactions (including severe pain, severe swelling, severe restriction of movement, persistent high fever, severe headache, or other systemic or local reactions) judged by the investigators.
* （6）Acute illness (acute illness refers to moderate or severe illness with or without fever) at the time of vaccination.
* （7）The axillary temperature >37.0℃ at the time of vaccination.

Ages: 42 Days to 77 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with serotype-specific pneumococcal IgG antibody concentration ≥ 0.35 ug/mL 30 days after primary vaccination | 30 days after primary vaccination
  Proportion of subjects with serotype-specific pneumococcal IgG antibody concentration ≥ 0.35 ug/mL 30 days after primary vaccination
Geometric mean concentration (GMC) of serotype-specific pneumococcal IgG antibody 30 days after primary vaccination | 30 days after primary vaccination
  Geometric mean concentration (GMC) of serotype-specific pneumococcal IgG antibody 30 days after primary vaccination

SECONDARY OUTCOMES:
Proportion of subjects with serotype-specific pneumococcal IgG antibody concentration ≥ 1.0 ug/mL 30 days after primary vaccination | 30 days after primary vaccination
  Proportion of subjects with serotype-specific pneumococcal IgG antibody concentration ≥ 1.0 ug/mL 30 days after primary vaccination
Geometric mean fold increase (GMI) of serotype-specific pneumococcal IgG antibody 30 days after primary vaccination | 30 days after primary vaccination
  Geometric mean fold increase (GMI) of serotype-specific pneumococcal IgG antibody 30 days after primary vaccination
Proportion of subjects with serotype-specific geometric mean titer measured by OPA ≥1:8 30 days after primary vaccination | 30 days after primary vaccination
  Proportion of subjects with serotype-specific geometric mean titer measured by OPA ≥1:8 30 days after primary vaccination
Geometric mean titer (GMT) of serotype-specific pneumococcal IgG antibody measured by OPA 30 days after primary vaccination | 30 days after primary vaccination
  Geometric mean titer (GMT) of serotype-specific pneumococcal IgG antibody measured by OPA 30 days after primary vaccination
Proportion of subjects with serotype-specific pneumococcal IgG antibody concentration ≥ 0.35 ug/mL 30 days after booster vaccination | 30 days after booster vaccination
  Proportion of subjects with serotype-specific pneumococcal IgG antibody concentration ≥ 0.35 ug/mL 30 days after booster vaccination
Proportion of subjects with serotype-specific pneumococcal IgG antibody concentration ≥ 1.0 ug/mL 30 days after booster vaccination | 30 days after booster vaccination
  Proportion of subjects with serotype-specific pneumococcal IgG antibody concentration ≥ 1.0 ug/mL 30 days after booster vaccination
Geometric mean concentration (GMC) of serotype-specific pneumococcal IgG antibody 30 days after booster vaccination | 30 days after booster vaccination
  Geometric mean concentration (GMC) of serotype-specific pneumococcal IgG antibody 30 days after booster vaccination
Proportion of subjects with serotype-specific geometric mean titer measured by OPA ≥1:8 30 days after booster vaccination | 30 days after booster vaccination
  Proportion of subjects with serotype-specific geometric mean titer measured by OPA ≥1:8 30 days after booster vaccination
Geometric mean titer (GMT) of serotype-specific pneumococcal IgG antibody measured by OPA 30 days after booster vaccination | 30 days after booster vaccination
  Geometric mean titer (GMT) of serotype-specific pneumococcal IgG antibody measured by OPA 30 days after booster vaccination
Incidence of adverse reactions (including systemic and local adverse reaction) 30 days after each dose of vaccination | 30 days after each dose of vaccination
  Incidence of adverse reactions (including systemic and local adverse reaction) 30 days after each dose of vaccination
Incidence of severe adverse event (SAE) within 6 months after the first doseof vaccination | 6 months after the first doseof vaccination
  Incidence of severe adverse event (SAE) within 6 months after the first doseof vaccination
Incidence of severe adverse event (SAE) 30 days after booster vaccination | 30 days after booster vaccination
  Incidence of severe adverse event (SAE) 30 days after booster vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Principal Investigator — Jiangsu Provincial Centre for Disease Control and Prevention
Locations (4):
- China (4):
  - Huaiyin District Center for Diseases Control and Prevention, Huai'an, Jiangsu
  - Hongze District Center for Disease Control and Prevention, Huai'an, Jiangsu
  - Lianshui County Center for Disease Control and Prevention, Huai'an, Jiangsu
  - Guanyun County Center for Disease Control and Prevention, Lianyungang, Jiangsu

REFERENCES:
- [Derived] Liang Q, Li H, Chang X, Zhang H, Hao H, Ye Q, Li G. A phase 3 clinical trial of MINHAI PCV13 in Chinese children aged from 7 months to 5 years old. Vaccine. 2021 Nov 16;39(47):6947-6955. doi: 10.1016/j.vaccine.2021.09.047. Epub 2021 Oct 24. PMID 34706841